CLINICAL TRIAL: NCT02506322
Title: Adjuvant Psychotherapy for Relapse Prevention in Early Adulthood (< 35 yr.) of Bipolar Disorder
Acronym: A2BipoLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Dresden (Other); University Hospital Goettingen (Other); Ludwig-Maximilians - University of Munich (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Bergmannsheil Bochum (Other); Charite University, Berlin, Germany (Other); Philipps University Marburg (Other); Goethe University (Other); Ruppiner Clinic, Psychiatric Clinic, Neuruppin (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Martin Hautzinger, University Professor of Clinical Psychology an Psychotherapy, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01EE1404C
Record Dates: First submitted 2014-12-19; First posted 2015-07-23 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder; Bipolar II Disorder; Relapse Prevention
MeSH Terms: conditions — Bipolar Disorder | interventions — MD1; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SEKT Cognitive-Behavioral-Emotional (Experimental): Specific psychotherapy (SEKT - 4 modules) for typical problems of Bipolar patients to maintain remission and to prevent relapse. Including classical elements of self observation, psychoeducation, cognitive and behavioral interventions, social rhythm but also emotion regulation and meta-cognitive techniques. Delivered in a group setting in 4 one day treatment workshops, each one month apart. Homework assignment and electronical monitoring during time between sessions.
  Interventions: Behavioral: SEKT - Cognitive-Behavioral-Emotional
- FEST Clinical Supportive Educational (Active Comparator): This supportive, active control psychotherapy (FEST) is using general principals and non-specific interventions such as positive attitude, optimism, support, empathy, focus on emotion, self-help, strengthening and eliciting own resources, time and room for discussion of personal experiences. Psychoeducation about illness and drug treatment (mood stabilizer) to facilitate compliance.
  Interventions: Behavioral: FEST - Clinical Supportive Educational

INTERVENTIONS:
Behavioral: SEKT - Cognitive-Behavioral-Emotional — This Bipolar Disorder specific psychotherapy has 4 modules:
  1. psychoeducation, life chart, relapse experiences, personalized explanation, early symptoms and recognition of a new episode, self observation
  2. Stress regulation, sleep-wake cycle, social rhythm, daily and weekly structure of life, life balance
  3. dysfunctional cognitions, cognitive techniques, meta-cognitive techniques, emotion regulation methods
  4. behavior changes, (social, problem solving) skill training, communication skills, crisis management
  Other Names: Specific Psychotherapy for Bipolar Disorder
  Arms: SEKT Cognitive-Behavioral-Emotional
Behavioral: FEST - Clinical Supportive Educational — This active control psychotherapy has 2 modules: (a) psychoeducation about Bipolar Disorder, the etiology and development of this disorder, drug options, effects and side effects of medication, compliance, how to handle unwanted side effects (b) group discussion and exchange about disorder relevant and personal relevant topics related to Bipolar Disorder, therapist is passive, encouraging, listening, verbalizing feelings and emotion, strengthening subjects resources
  Other Names: Supportive, non-specific psychotherapy for Bipolar Disorder
  Arms: FEST Clinical Supportive Educational

SUMMARY:
This efficacy study compares an adjuvant specific psychotherapy and an active control intervention for Bipolar Disorder under mood stabilizer to prevent relapse an maintain remission. Patients should be in their early (18-30 yr.) phase of illness without having suffered of to many affective episodes (below 6), already. In addition, psychological, social, and neurobiological mediators and moderators well be identified.

DETAILED DESCRIPTION:
There is still a lack of controlled outcome and follow-up studies about the role of adjuvant psychotherapy in Bipolar Disorder. By treating older subjects having suffered of multiple affective episodes, the potential benefit of psychotherapy to prevent relapse and help to adjust to this chronic illness might be underestimated. In addition, the investigators have no knowledge of mechanism (mediators) of positive changes by successful psychotherapy and of subjects with good outcome of adjuvant psychotherapy (moderators, indicators, predictors). Possible mediators and moderators can be sociodemographic, psychological (cognitive, interactional), and/or biological (neuronal, genetic). The planned study will address all three areas of questions. In a multi-center study, 300 younger subjects suffering of a Bipolar Disorder will be included and provide with one of two treatments in addition to stable medication. Moderators and mediators are selected on promising preliminary results and based on a psycho-biological understanding of Bipolar Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and Bipolar II Disorder,
* 18 to 55 years of age,
* giving informed consent to assessment, treatment, and randomization,
* currently remitted (for at least 4 weeks) and taking medication,
* less than 6 previous affective episodes

Exclusion Criteria:

* currently symptomatic (depressed, manic, hypomanic),
* suicidal,
* not taking medication,
* schizo-affective, schizophrenic, borderline personality disorder,
* not giving or withdrawing consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Time to new affective episode | 18 months
  At baseline, subjects have to be remitted. Psychotherapies focus on maintenance and relapse prevention. Relapse will be assessed by LIFE interview every six month

SECONDARY OUTCOMES:
Qick-Inventory of Depressive Symptoms | 18 months
  Clinician ratings of depressive symptoms
Social functioning | 18 months
  Clinician rating social functioning (GAF)
Neurobiological changes (functional, genetic) (functional MRI) | 6 months
  functional MRI at baseline and after six month
Young Mania Rating Scale | 18 months
  Clinician ratings of manic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Martin HAUTZINGER, PhD, Principal Investigator — Department Psychology University Tuebingen
Locations (1):
- Eberhard Karls University, Tübingen, Germany

REFERENCES:
- [Background] Meyer TD, Hautzinger M. Cognitive behaviour therapy and supportive therapy for bipolar disorders: relapse rates for treatment period and 2-year follow-up. Psychol Med. 2012 Jul;42(7):1429-39. doi: 10.1017/S0033291711002522. Epub 2011 Nov 21. PMID 22099722
- [Derived] Hautzinger M; A2 BipoLife Consortium. Adjuvant Psychotherapies to Prevent Relapse in Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Sep 1;81(9):855-862. doi: 10.1001/jamapsychiatry.2024.1310. PMID 38837133
- [Derived] Meyer K, Hindi Attar C, Fiebig J, Stamm T, Bassett TR, Bauer M, Dannlowski U, Ethofer T, Falkenberg I, Jansen A, Juckel G, Kircher T, Mulert C, Leicht G, Rau A, Ritter D, Ritter P, Trost S, Vogelbacher C, Walter H, Wolter S, Hautzinger M, Bermpohl F. Boosting the Theory of Mind Network: Specific Psychotherapy Increases Neural Correlates of Affective Theory of Mind in Euthymic Bipolar Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 May;8(5):572-580. doi: 10.1016/j.bpsc.2022.08.013. Epub 2022 Sep 8. PMID 36087699
- [Derived] Stamm TJ, Zwick JC, O'Malley G, Sondergeld LM, Hautzinger M. Adjuvant psychotherapy in early-stage bipolar disorder: study protocol for a randomized controlled trial. Trials. 2020 Oct 13;21(1):845. doi: 10.1186/s13063-020-04755-8. PMID 33050952